CLINICAL TRIAL: NCT04967742
Title: A Phase I, Open-Label Extension Study to Evaluate the Safety, Tolerability, and Immunogenicity of UB-612 Vaccine in Healthy Adult Volunteers
Brief Title: A Extension Study to Evaluate the Safety, Tolerability, and Immunogenicity of UB-612 COVID-19 Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United Biomedical Inc., Asia (Industry)
Collaborators: Vaxxinity, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V-123
Record Dates: First submitted 2021-07-12; First posted 2021-07-20 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — UB-612 COVID-19 vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A group: 1 booster dose of UB-612 vaccine 100 μg (Experimental): 1 booster dose for subjects at UB-612 vaccine 10 μg in V-122 study.
  Interventions: Biological: UB-612
- B group: 1 booster dose of UB-612 vaccine 100 μg (Experimental): 1 booster dose for subjects at UB-612 vaccine 30 μg in V-122 study.
  Interventions: Biological: UB-612
- C group: 1 booster dose of UB-612 vaccine 100 μg (Experimental): 1 booster dose for subjects at UB-612 vaccine 100 μg in V-122 study.
  Interventions: Biological: UB-612

INTERVENTIONS:
Biological: UB-612 — UB-612 includes a designer S1-RBD-sFc fusion protein formulated with designer Th and CTL epitope peptides selected from immunodominant M, S2 and N regions known to bind to human MHC I and II.

SUMMARY:
This is an extension study to evaluate the safety, tolerability and immunogenicity of one booster dose of UB-612 COVID-19 vaccine in adults who completed two vaccinations of UB-612 vaccine 10, 30, and 100 μg in V-122 study.

DETAILED DESCRIPTION:
This is an extension study to evaluate the safety, tolerability and immunogenicity of one booster dose of UB-612 COVID-19 vaccine in adults who completed two vaccinations of UB-612 vaccine 10, 30, and 100 μg in V-122 study. 60 subjects will receive one booster dose of UB-612 vaccines 100 μg with the same dose which was offered in Phase II study, at least 6 months after first vaccination. In this study, there will be 3 clinical visits. Subjects will come to the clinics at Day 1, Day 15, and Day 85.

ELIGIBILITY:
* Inclusion Criteria

  1. Male or non-pregnant female who previously participated in and completed two vaccinations in the V-122 Study.
  2. Women of childbearing potential and men must agree to practice medically effective contraception during study period.
  3. Able to understand the content and possible risks of informed consent and willing to sign the Informed Consent Form (ICF).
  4. Able to understand and agrees to comply with all study procedures and be available for all study visits.
  5. Ear temperature ≤ 38.0°C.
  6. At screening visit, at least 6 months after first vaccination in the V-122 study.
* Exclusion Criteria

  1. Female who is pregnant or positive in pregnancy test at screening visit.
  2. Female who is breast-feeding or plans to breastfeed within 90 days after booster vaccination.
  3. Any acute illness, as determined by the study investigator 3 days before booster vaccination.
  4. Prior administration of attenuated, nucleic acid (mRNA or DNA) or vectored vaccines in last 1 month before booster vaccination or expectation of such vaccines in the month after booster vaccination.
  5. Prior administration of subunit vaccine or inactivated vaccine in last 14 days before booster vaccination or expectation of receipt of such vaccines in the 14 days after booster vaccination.
  6. Any medical disease or condition that, in the opinion of the study investigator, may confound the results of the study or pose an additional risk to the subjects by their participation in the study.
  7. Previous exposure to SARS-CoV-2 or receipt of an investigational or EUA vaccine product for the prevention of COVID-19, MERS or SARS except UB-612.
  8. Subjects who take part in another clinical study, other than V-122 study, within 12 weeks prior to the day of informed consent.
  9. Prior administration of immunoglobulins and/or any blood products in last 4 months before booster vaccination.
  10. Prior chronic administration of immunosuppressant or corticosteroids, cytotoxic treatment in last 6 months before first vaccination.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2021-08-22 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
GMT of neutralizing antibody against SARS-CoV-2 | Day 1
  Evaluation of Immunogenicity
GMT of neutralizing antibody against SARS-CoV-2 | Day 15
  Evaluation of Immunogenicity
GMT of neutralizing antibody against SARS-CoV-2 | Day 85
  Evaluation of Immunogenicity
Geometric mean fold increase of neutralizing antibody against SARS-CoV-2 | Day 15
  Evaluation of Immunogenicity
Geometric mean fold increase of neutralizing antibody against SARS-CoV-2 | Day 85
  Evaluation of Immunogenicity
Occurrence of adverse reactions and the percentage of subjects with ≥ Grade 3 adverse events | Within 7 days after vaccination
  Evaluation of Safety

SECONDARY OUTCOMES:
GMT of antigen-specific antibody (Anti-S1-RBD) | Day 1
  Evaluation of Immunogenicity
GMT of antigen-specific antibody (Anti-S1-RBD) | Day 15
  Evaluation of Immunogenicity
GMT of antigen-specific antibody (Anti-S1-RBD) | Day 85
  Evaluation of Immunogenicity
Geometric mean fold increase of antigen-specific antibody (Anti-S1-RBD) | Day 15
  Evaluation of Immunogenicity
Geometric mean fold increase of antigen-specific antibody (Anti-S1-RBD) | Day 85
  Evaluation of Immunogenicity
Correlation between the immune response detected by ELISA and live virus neutralization test | During the study period
  Evaluation of Immunogenicity
Occurrence of SAEs, AESIs, MAAEs and SAEs | During the study period
  Evaluation of Safety

OTHER OUTCOMES:
T cell responses to UB-612 COVID-19 Vaccine | Day 1
  Evaluation of Immunogenicity
T cell responses to UB-612 COVID-19 Vaccine | Day 15
  Evaluation of Immunogenicity
T cell responses to UB-612 COVID-19 Vaccine | Day 85
  Evaluation of Immunogenicity
GMT of neutralizing antibody against SARS-CoV-2 variants | Day 1
  Evaluation of Immunogenicity
GMT of neutralizing antibody against SARS-CoV-2 variants | Day 15
  Evaluation of Immunogenicity
GMT of neutralizing antibody against SARS-CoV-2 variants | Day 85
  Evaluation of Immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Yi Wang, Ph.D, Study Chair — United Biomedical Inc., Asia
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Wang CY, Hwang KP, Kuo HK, Peng WJ, Shen YH, Kuo BS, Huang JH, Liu H, Ho YH, Lin F, Ding S, Liu Z, Wu HT, Huang CT, Lee YJ, Liu MC, Yang YC, Lu PL, Tsai HC, Lee CH, Shi ZY, Liu CE, Liao CH, Chang FY, Chen HC, Wang FD, Hou KL, Cheng J, Wang MS, Yang YT, Chiu HC, Jiang MH, Shih HY, Shen HY, Chang PY, Lan YR, Chen CT, Lin YL, Liang JJ, Liao CC, Chou YC, Morris MK, Hanson CV, Guirakhoo F, Hellerstein M, Yu HJ, King CC, Kemp T, Heppner DG, Monath TP. A multitope SARS-CoV-2 vaccine provides long-lasting B cell and T cell immunity against Delta and Omicron variants. J Clin Invest. 2022 May 16;132(10):e157707. doi: 10.1172/JCI157707. PMID 35316221